CLINICAL TRIAL: NCT06133192
Title: A Multi-center Randomized Phase II Study Comparing Corticosteroids Alone Versus Corticosteroids and Extracorporeal Photopheresis as First-line Treatment of Grade II Acute Graft-versus-host Disease With Skin Involvement Occuring After Allogeneic Stem Cell Transplantation
Brief Title: Steroids Versus ECP and Steroids as First-line Treatment of Grade II Acute GVHD
Acronym: COPAVEHDI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Marie-Thérèse RUBIO, PU-PH, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-508614-41-00
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Methoxsalen; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroids alone (Active Comparator): Steroids 2 mg/kg/day
  Interventions: Drug: Steroids
- ECP + steroids (Experimental): Steroids 2 mg/kg abd ECP x 2 per week for 1 months and once a week for 2 months
  Interventions: Drug: Uvadex

INTERVENTIONS:
Drug: Uvadex — Uvadex use for ECP
  Arms: ECP + steroids
Drug: Steroids — steroids 2 mg/kg/d
  Arms: Steroids alone

SUMMARY:
The goal of this clinical trial is to compare as a first line of grade II skin acute GVHD sconventional treatment with steroids alone to a combination of steroids and extracoporeal photopheresis (ECP)

The primary end point will compare Freedom from treatment failure at 6 months from randomization as defined by meeting all the following 4 conditions:

* to be alive
* without relapse of the hematological disease
* without having required a new line of treatment for acute GVHD
* without initiating a systemic treatment for chronic GVHD.

DETAILED DESCRIPTION:
A multi-center randomized phase II study comparing corticosteroids alone (standard of care) versus corticosteroids and extracorporeal photopheresis as first-line treatment of Grade II acute graft-versus-host disease with skin +/- upper gastrointestinal involvement occurring after allogeneic stem cell transplantation

Corticosteroids will be started at 2 mg/kg in both arms and will be tapered once acute GVHD achieves complete remission according to strict protocol guidelines (-20% of the daily dose per week until 1 mg/kg and then 10 mg twice a day in order to stop steroids within 2 to 3 months from randomization).

Extracorporeal Photopheresis (ECP) will be performed in the experimental arm : 2 sessions/week during 4 weeks then 1 session/week during 8 weeks), i.e. a total of 16 ECP sessions in 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* allogeneic hematopoietic stem cell transplantation received (from any type of graft and donor) after malignant or non malignant disease
* patient suffering from Grade II acute GVHD with skin +/- high GI involvement (stage 2-3 skin + upper gastrointestinal tract or skin stage 3) in the 3 months following stem cell transplantation
* patient requiring first line treatment for acute GVHD
* patient able to start PCE therapy in the 3 days after randomization
* validation of the presence of a peripheral or central venous access (its type should be conform to the recommendations described in the Therakos Cellex operator manual), allowing to perform PCE sessions weekly during 3 months. In the absence of appropriate preexisting central line at inclusion, peripheral access will be preferred.
* leukocytes > 1.5 G/l, platelets > 30 G/l, hematocrit > 27% (blood transfusion are permitted), based on the last available blood testing results,
* patient with French Health Insurance,
* patient informed about the clinical trial content and organization,
* informed consent form signed.

Exclusion Criteria:

* - Grade 1 acute GVHD,
* acute GVH grade > II or acute GVH with lower gastrointestinal tract or with liver involvement,
* relapse of the hematologic disease at time of acute GVHD,
* uncontrolled ongoing infection at time of inclusion: bacterial or fungal infections, CMV reactivation with increasing CMV viral load,
* HIV positivity or replicative HBV or HCV infection (based on pre-transplant assessment),
* patient with allergy or contraindications to UVADEX, extracorporeal photopheresis, steroids, or posaconazole (see details in the study protocol),
* woman of childbearing age without efficient contraceptive method, pregnancy or breast feeding woman,
* patient with history of profound venous thrombosis in the last 5 years,
* patient included in another acute GVHD prospective clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from treatment failure | at 6 months from randomization
  To be alive, without disease relapse, without second line treatment for acute GVHD and without systemic treatment for chronic GVHD

SECONDARY OUTCOMES:
steroid cumulative dose | at 6 months from randomization
  cumulative dose of steroids over time
infections | at 6 months from randomization
  incidence rate of infections (bacteremia, septicemia, fungal infections, parasite and virus
chronic GVHD | at 12 months from randomization
  incidence and severity of chronic GVHD
non-relapse mortality | at 12 months from randomization
  non-relapse mortality rate
relapse | at 12 months from randomization
  incidence of disease relapse
overall survival | at 12 months from randomization
  overall survival logrank

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No